CLINICAL TRIAL: NCT04999371
Title: Effects of Training Combined With a Small Financial Incentive on Reducing Alcohol Consumption: Study Protocol for a Cluster-randomized Controlled Trial
Brief Title: Effects of Training Combined With a Small Financial Incentive on Reducing Alcohol Consumption
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Yu Sun, Ph.D., Assistant Director, PKU China Center for Health Economic Research (CCHER)Yu Sun, Ph.D. Assistant Director, PKU China Center for Health Economic Research (CCHER), Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ccher_liangshan alcohol
Record Dates: First submitted 2021-07-24; First posted 2021-08-10 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Ethanol; Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control without intervention (No Intervention): No information or cash incentives are provided to the participants in the control group, but it is also necessary to collect the information of the participants in the control group and perform an alcohol test. Therefore, the project team will provide a certain degree of compensation for participants in the control group (participants of the intervention group also will receive this part of compensation).
- Mobile-based information intervention (Active Comparator): The participants in this group received free three-time counsel and constant multi-media messages about the topic of alcohol consumption for three months. One-to-one counseling services will be provided via a telephone call, which is based on World Health Organization (WHO) recommendations. A total of three counsels are conducted, which are set on the second week, sixth and tenth week after the baseline survey.
  Interventions: Behavioral: Brief Alcohol Intervention
- Mobile-based information intervention with performance-based incentive (Active Comparator): The participants in this group were conducted by deducting money. Firstly, a certain amount of vouchers were given to the participants, which was equivalent to the reward for passing seven tests. Then, the voucher would be deducted according to every test result. Finally, the participants will receive cash according to the vouchers.
  Interventions: Behavioral: Brief Alcohol Intervention; Behavioral: Financial Incentive Intervention

INTERVENTIONS:
Behavioral: Brief Alcohol Intervention — The participants in the treatment group received free three-time counsel and constant multi-media messages about the topic of alcohol consumption for three months. One-to-one counseling services will be provided via a telephone call, which is based on World Health Organization (WHO) recommendations. A total of three counsels are conducted, which are set on the second week, sixth and tenth week after the baseline survey.
  Brief intervention counselors are from the team of this study and trained by Hongkong University. All counselors are required to attend a full-day workshop before participant recruitment. The contents of the workshop include (1) knowledge of excessive drinking harms and benefits of controlling drinking; (2) overview of AUDIT; (3) alcohol reduction advice; (4) a standard procedure of brief intervention.
  Arms: Mobile-based information intervention; Mobile-based information intervention with performance-based incentive
Behavioral: Financial Incentive Intervention — The participants in financial Incentive intervention group were conducted by deducting money. Firstly, a certain amount of vouchers were given to the participants, which was equivalent to the reward for passing seven tests. Then, the voucher would be deducted according to every test result. Finally, the participants will receive cash according to the vouchers.
  Arms: Mobile-based information intervention with performance-based incentive

SUMMARY:
The existing alcohol intervention studies are mainly conducted in developed countries, few studies have focused on alcohol consumption among ethnic minority migrant people in developing countries. To address this gap, the investigators aim to evaluate the effects of a brief intervention combined with a small financial incentive on alcohol consumption and health outcomes among the migrated population in Liangshan Prefecture. This study was conducted in Liangshan Prefecture for two reasons: first, Liangshan is a region located in the southwestern of Sichuan province and is populated by Yi minority, and the average income in Liangshan is just about two-thirds of the national average income. Second, a study found that the drinking rate of the Yi minority (47.9%) is higher than that of other regions in China.

The aim of this paper is to provide an overview of alcohol consumption among the ethnic populations in China and to test the feasibility and efficacy of small financial incentives with brief advice intervention targeting the reduction of harmful drinking behaviors among poor people.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Age<18 and Age>65
* Scores of AUDIT<8
* Do not speak mandarin
* Less than three-months residence at Xichang
* Income not calculated by hour wage or piece-rate wage
* Those who have previous abstinence experience, epilepsy, liver disease, and is using sedative drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 443 (Estimated)
Dates: Start 2021-07-29 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Self-reported drinking quantity | 3 months
  (drinks per week)
Self-reported binge drinking frequency | 3 months
  (number of binges per week)
Self-reported drinking frequency. | 3 months
  (drinking days per week)
Self-reported drinking intensity. | 3 months
  (number of drinks per drinking day)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University China Center for Health Economic Research, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The data can be provided according to the needs of the researcher, but does not include all personal data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available in 2024
Access Criteria: The data are for research purposes only

REFERENCES:
- [Derived] Li S, Wu Z, Liu S, Sun Y, Liu GG. Effect of a brief intervention with small financial incentives on alcohol consumption in China: study protocol for a randomised controlled trial. BMJ Open. 2022 May 18;12(5):e056550. doi: 10.1136/bmjopen-2021-056550. PMID 35584882